CLINICAL TRIAL: NCT03856359
Title: Pilot, Single Center, Open, Trial of Rifaximin in Probable Alzheimer's Disease
Brief Title: Trial of Rifaximin in Probable Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00093318
Record Dates: First submitted 2019-01-31; First posted 2019-02-27 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rifaximin (Experimental): rifaximin 550 milligrams (mg) orally twice daily for 3 months
  Interventions: Drug: Rifaximin 550 milligrams (MG)

INTERVENTIONS:
Drug: Rifaximin 550 milligrams (MG) — Rifaximin (Xifaxan, Salix Pharmaceuticals, Bridgewater, N.J.) (See Package Insert) is a drug that is approved by the FDA for use in humans for the treatment of Hepatic Encephalopathy, Traveler's Diarrhea and Irritable Bowel Syndrome. It is commercially available. It will be used in accordance with approved labeling as pertains to dosage and administration for Hepatic Encephalopathy, contraindications and warnings. However, it will be used investigationally in this trial as rifaximin is not FDA approved for the treatment of Alzheimer's Disease.

SUMMARY:
This study aims to improve cognition and function in patients with Alzheimer's Disease (AD) by administering the oral antibiotic, Rifaximin.

Rifaximin is a virtually non-absorbed antibiotic with the unique properties of lowering blood ammonia levels and altering gut microbiota. It is FDA approved for use in patients with hepatic encephalopathy. Rifaximin lowers blood ammonia by altering fecal flora by blocking bacterial RNA synthesis and also by increasing small bowel glutaminase. The Investigators hypothesize that rifaximin will improve cognition and function in AD patients by lowering blood ammonia and / or lowering circulatory pro-inflammatory cytokines secreted by harmful gut bacteria. The Investigators will enroll up to 10 subjects with probable middle stage Alzheimer's Disease. The subjects will be given rifaximin 550 mg orally twice daily for 3 months after evaluation to ensure they have no contraindications. Physician clinical and safety assessments, adverse events, as well as the ADAS-Cog-11 will be administered at baseline and at the 3 month endpoint and two months after stopping treatment (at month 5). Interim safety checks will occur via phone calls one week after baseline and then every 2 weeks till end point. Serum neuronal biomarkers, ammonia levels and pro-inflammatory and anti-inflammatory compounds will also be measured at those times. Bodily fluids (Stool samples) will also be collected. Because of a small risk of developing C. difficile up to 2 months following the last administration of rifaximin, the subjects will be followed for an additional 2 months after the 3 month treatment ends.

Rifaximin is contraindicated in patients with hypersensitivity to rifaximin or rifamycin antimicrobials. Hypersensitivity reactions include exfoliative dermatitis, angioneurotic edema, and anaphylaxis. Clostridium difficile associated diarrhea is a risk whenever a patient is maintained chronically on antibiotics, with complications ranging from mild diarrhea to fatal colitis. Drug resistant bacteria can also result from long term use. There is increased systemic exposure to rifaximin in patients with severe hepatic impairment or in patients who are taking P-glycoprotein inhibitors concomitantly. Regarding use in geriatric patients, there were no reported overall differences in the safety of the drug when used in patients 65 years of age or over, when compared with younger subjects.

DETAILED DESCRIPTION:
This study aims to improve cognition and function in patients with Alzheimer's Disease (AD) by administering the oral antibiotic, rifaximin. Rifaximin is a virtually non-absorbed antibiotic with the unique properties of altering gut microbiota and lowering blood ammonia levels. It is FDA approved for use in patients with hepatic encephalopathy. Rifaximin lowers blood ammonia by blocking gut bacterial RNA synthesis and also by increasing small bowel glutaminase. The Investigators hypothesize that rifaximin will improve cognition and function in AD patients by mechanisms such as lowering circulatory pro-inflammatory cytokines secreted by harmful gut bacteria or lowering blood ammonia.

Rifaximin is a relatively gut-specific antibiotic that interferes with by binding to the transcription subunit of bacterial . Because Rifaximin is absorbed poorly, most of the drug taken RNA polymerase orally stays in the gastrointestinal tract. It has been available since 2004 in the US and has orphan gastrointestinal tract drug status for hepatic encepalopathy. Rifaximin's relatively good safety profile and its ability to alter gut flora and lower blood ammonia have made it an attractive drug to treat hepatic encephalopathy or conditions such as traveller's diarrhea. The Investigators hypothesize that rifaximin will improve cognition and function in AD patients by mechanisms such as lowering circulatory pro-inflammatory cytokines secreted by harmful gut bacteria or lowering blood ammonia.

The Investigators will measure a variety of blood markers, such as pro-inflammatory and anti-inflammatory compounds, and analyze fecal microbiota in patients with AD before and after 3 months of rifaximin therapy. If patients exhibit measurable improvement in cognition and function, The Investigators will analyze our data to see if their improvement correlates with a shift towards anti-inflammatory species in the gut and a similar shift in the blood cytokine panel to favoring anti-inflammatory compounds.

Evidence supporting our hypothesis for this study is presented below.

Gut Microbiota Dysbiosis

The gut harbors 95% of the total human microbiome and is made up of more than 5,000 taxa. Gut species remain relatively constant throughout adulthood until the seventh decade, when it becomes less diverse, harboring higher numbers of Proteobacteria and lower numbers of Bifidobacteria. An imbalance in the gut bacterial species can weaken the intestinal barrier and create system wide inflammation via gut lymphoid tissue which comprises 70% - 80% of the immune system. Blood brain barrier permeability is also altered. The gut bacteria secrete pro-inflammatory compounds and neuroactive molecules that include serotonin, gamma-aminobutyric acid (GABA), catecholamines and acetylcholine which cross the blood brain barrier and cause brain inflammation and brain dysfunction.

A growing number of pro-inflammatory compounds secreted by gut bacteria and seen in patients with AD are being discovered. These include interleukin (IL) - 6, tumor necrosis - alpha and the inflammasome complex (NLRP3). A recent study revealed higher numbers of Escherichia and Shigella in the gut of amyloid positive AD patients when compared with healthy controls and this correlated with higher levels of circulating pro-inflammatory cytokines. The AD patients also had lower numbers of gut Eubacterium rectale and this correlated with lower levels of circulating anti-inflammatory compounds than seen in controls. Other researchers found that a preponderance of gut Bacteroides and Blautia and reduced numbers of SMB53 and Dialister correlated with elevated levels of brain amyloid Cerebrospinal Fluid (CSF) biomarkers. Interestingly, Clostridium tyrobutyricum and Bacteroides thetaiotaomicron, have been shown to actually increase the integrity of the blood brain barrier by enhancing expression of tight junction proteins and helping to maintain brain homeostasis. Recent evidence also suggests that neurotransmitters and neuropeptides secreted by bacteria in the gut activate vagal nerve ascending fibers, influencing brain function.

Ammonia Neurotoxicity

A second theory is that the blood brain barrier allows greater amounts of ammonia into the AD brain, triggering or worsening pre-existent changes. The possibility that ammonia is at least partly responsible for the pathologic changes seen in the AD brain was first proposed by Seiler in 1993, when he noted that some of the changes in the AD brain can also be seen in the brains of hyperammonemic patients. Arteriovenous sampling in early stage normoammonemic AD patients demonstrated higher endogenous cortical ammonia compared to young control subjects Low glutamine synthetase levels have been found to correlate with increased density of amyloid deposits in the AD brain.

The brain also receives exogenous ammonia, of which the gut is a major source. The aging colon contains a greater percentage of protein fermenting bacteria than is seen in the colon of younger patients.

Rifaximin lowers blood ammonia by altering fecal flora by blocking bacterial RNA synthesis and also by increasing small bowel glutaminase.

The Investigators hypothesize that Rifaximin will improve cognition and function in AD patients by lowering circulatory pro-inflammatory cytokines secreted by harmful gut bacteria and / or lowering blood ammonia levels. The subjects will be given rifaximin 550 mg orally twice daily for 3 months after evaluation to ensure they have no contraindications. Physician clinical and safety assessments, adverse events, as well as the ADAS-Cog11 will be administered at baseline and at the 3 month endpoint. Interim safety checks will occur via phone calls one week after baseline and then every 2 weeks till 3 month end point. Serum neuronal biomarkers, ammonia levels and pro-inflammatory and antiinflammatory compounds will also be measured at those times. Bodily fluids (Stool samples) will also be collected. Because of a small risk of developing C. difficile up to 2 months following the last administration of rifaximin, the subjects will be followed for an additional 2 months after the 3 month treatment ends.

This is an open label pilot study designed to provide preliminary evidence on the clinical efficacy of rifaximin in improving cognition in AD patients. The Investigators will be looking for improvement in test scores and changes in serum levels of neuronal markers, circulating cytokine pro-inflammatory compounds and colonic microbiota following treatment. The Investigators will also be collecting data regarding the safety of long term use of this non-absorbed antibiotic for this disease. This pilot may form the basis for a future larger randomized, double blind controlled study to further test this hypothesis.

The rifaximin dosage and route of administration are the same as that used to treat hepatic encephalopathy, for which the drug and dosage are FDA approved. The dose will remain the same throughout the 3 month study of rifaximin administration unless stopped for safety reasons. The age and study sample of mild to moderate probable AD is similar to that used in AD prior trials. The Investigators will select our sample to be medically stable and free of hepatic disease and not having had recent antibiotic therapy to minimize risk for C Difficile infection.

The end of the study will occur 5 months after baseline testing and first administration of the drug. While drug administration will conclude and endpoint testing will be done at 3 months, The Investigators will continue to follow each subject for an additional 2 months, as C. difficile infectious diarrhea can occur up until 2 months after stopping an antibiotic.

ELIGIBILITY:
Inclusion Criteria:

* · Probable Alzheimer's Disease (National Institute of Neurological Disorders and Stroke (NINDS) criteria), mild to moderate severity

  * Ages 55-85; both genders
  * Mini Mental State Exam (MMSE) scores 10-23
  * Willing and able to comply with all scheduled clinic visits.
  * Stable medical health
  * Has a family or professional caregiver who has regular contact with subject
  * Ability to consent or legal guardian who can consent
  * Living at home or in a facility
  * On no AD therapies or on stable (2 months) concurrent AD therapies

Exclusion Criteria:

* Past history of C diff infection
* Assessment, laboratory examination, physical examination or any other medical condition or circumstance making the volunteer unsuitable for participation in the study in the judgment of the study clinicians
* Allergy to Rifaximin
* Antibiotic use or hospitalization in the last 6 months
* Are taking medications that interact with rifaximin and/or pose a safety risk in the judgment of the PI
* Clinically significant abnormal hepatic or renal function
* Uncorrected thyroid or B12 abnormalities
* Participation in another investigational drug trial in the past 30 days
* History of febrile illness within 5 days prior to the study period
* Known Hyperammonemia caused by:

Valproic acid Chemotherapy Lung transplant Bariatric surgery Ureterosigmoidoscopy Hyperalimentation Urinary tract infection Errors of metabolism: urea cycle, enzyme deficiencies, organic acidemias, fatty acid oxidation, amino acid transport defects

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Suhocki, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from referrals and the community via advertisement. Subjects and caregivers compensated for participation in the study to cover travel and time.
Period: Overall Study
Arm/Group | Rifaximin
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 72 [50 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Diarrhea Caused by Clostridium Difficile
Description: Collected at every visit and follow-up phone visits. A rare side effect of Rifaximin is diarrhea caused by clostridium difficile. This is a very serious form of diarrhea that can be fatal if not treated. The investigators will be following the patients closely during treatment and for 2 months following treatment to see if the patient has any signs or symptoms of this diarrhea. If a patient does develop clostridium difficile diarrhea, they will be promptly treated.
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
Participants | 5

2. Primary Outcome: Change in ADAS Cog 11 Scores
Description: Change in Alzheimer's Disease Assessment Scale - Cognition test with 11 tasks (ADAS Cog 11) scores following 3 months of oral Rifaximin. Scores range from minimum 0 - maximum 70. Higher scores mean worse outcome.
Time Frame: At baseline and at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
score on a scale | 30.5 [30.3 to 31]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.60, t-test, 2 sided

3. Secondary Outcome: Change in Tolerability as Measured by Number of Adverse Events (AE).
Description: Assessed at every visit. The patients will be followed closely to see if they are tolerating the drug, Rifaximin. The of the number of side effects would indicate that the patient may not be tolerating the drug. Most of these side effects are minor and include headache, nausea, vomiting, tiredness. A potentially fatal side effect would be the development of clostridium difficile diarrhea. The investigators will be following the patients closely during treatment and for 2 months following treatment to see if the patient has any signs or symptoms of this diarrhea. If a patient does develop clostridium difficile diarrhea, they will be promptly treated.
Time Frame: Baseline, 3 months, 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
Participants | 7

4. Secondary Outcome: Change in Cognitive Performance on the Mini-Mental State Exam (MMSE)
Description: Change from baseline global cognitive scores at month 3). Global cognitive performance will be assessed by a psychometrician using the (MMSE). It is a brief cognitive questionnaire with a maximum score of 30 points. MMSE range is 0-30 with lower scores indicating worse performance. The number of correct answers is added to generate the total score.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
score on a scale | -0.3 [-1.8 to 1.2]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.67, t-test, 2 sided

5. Secondary Outcome: Participants With Treatment Emergent Adverse Events as Reported by the Subject That Required a Change in Safety Measures
Description: Emergent AEs that required a change in safety measures. These were AEs that were found when talking to or examining the subjects.
Time Frame: Safety will be measured through adverse events throughout study, at month 3 and by phone call at month 5 (2 months after treatment termination).
Measure: Number; unit: percentage of participants
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
percentage of participants | 0

6. Secondary Outcome: Changes From Baseline in Ammonia Level
Description: Change in ammonia levels following treatment with Rifaximin.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
mg/dL | 0.1 [-7.06 to 7.25]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.73, t-test, 2 sided

7. Secondary Outcome: Development of Clostridium Difficile Diarrhea
Description: Observing for development of diarrhea due to Clostridium difficile
Time Frame: Baseline to 3 months
Measure: Number; unit: percentage of subjects
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
percentage of subjects | 0

8. Secondary Outcome: Total Tau
Description: Change in serum Total tau after 3 months Rifaximin administration.
Time Frame: Baseline, 3 months
Measure: Number (95% Confidence Interval); unit: ng/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
ng/mL | -0.17 [-0.61 to 0.26]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.38, t-test, 2 sided

9. Secondary Outcome: Phosphorylated Tau
Description: Change in Phosphorylated tau following 3 months oral Rifaximin
Time Frame: at baseline and at 3 months
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
ng/mL | -0.39 [-1.07 to 0.30]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.23, t-test, 2 sided

10. Secondary Outcome: Change in Glial Fibrillary Acidic Protein (GFAP)
Description: Change in Glial Fibrillary Acidic Protein (GFAP) after 3 months of oral Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -39.76 [-99.46 to 19.93]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.17, t-test, 2 sided

11. Secondary Outcome: Change in Neurofilament Light (Nfl) Levels
Description: Change in Neurofilament Light levels after Rifaximin for 3 months
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: ng/L
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
ng/L | -4.22 [-6.71 to -1.72]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.004, t-test, 2 sided

12. Secondary Outcome: Change in Interleukin 10 (IL-10)
Description: Change in Interleukin 10 following 3 months Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | 00.70 [-4.85 to 3.46]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.7, t-test, 2 sided

13. Secondary Outcome: Changes in Interleukin 13 (IL-13) Following Treatment With Rifaximin
Description: Interleukin 13 levels after Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -1.78 [-3.9 to 0.33]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.09, t-test, 2 sided

14. Secondary Outcome: Change in Interleukin 1B (IL-1B)
Description: Change in Interleukin 1B following Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -0.1 [-2.06 to 1.87]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.65, t-test, 2 sided

15. Secondary Outcome: Change in Interleukin 2 (IL-2)
Description: Change in Interleukin 2 following Rifaximin
Time Frame: Baseline, 3 months
Population: 10 patients with Alzheimer's Disease
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -0.33 [-0.93 to 0.27]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.18, t-test, 2 sided

16. Secondary Outcome: Change in Interleukin 4 (IL-4)
Description: Change in Interleukin 4 after Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -17.40 [-68.73 to 33.93]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.44, t-test, 2 sided

17. Secondary Outcome: Change in Interleukin 5 (IL-5)
Description: Change in Interleukin 5 after Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -0.87 [-2.34 to 0.60]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.20, t-test, 2 sided

18. Secondary Outcome: Change in Interleukin 8 (IL-8)
Description: Change in Interleukin 8 after Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -1.31 [-5.81 to 3.20]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.53, t-test, 2 sided

19. Secondary Outcome: Change in Interleukin 6 (IL-6)
Description: Change in Interleukin 6 following Rifaximin
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -1.62 [-3.39 to 0.15]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.07, t-test, 2 sided

20. Secondary Outcome: Change in Tumor Necrosis Factor a
Description: Change in Tumor Necrosis Factor a
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rifaximin
Number analyzed (Participants) | 10
pg/mL | -0.46 [-1.55 to 0.64]
Statistical Analysis 1: Comparison: Rifaximin; Test type: Superiority; p = 0.36, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | Rifaximin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=10)
Decline in cognitive ability (Nervous system disorders) | 1 (1)
Increased confusion (Nervous system disorders) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Hand tremor (Nervous system disorders) | 1 (1)
Fell out of chair (Musculoskeletal and connective tissue disorders) | 1 (1)
Fell (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03856359/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03856359/SAP_001.pdf
  • Informed Consent Form (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03856359/ICF_002.pdf